## Effects of Moringa Oleifera and Royal Jelly Supplementation on Nutritional Status and Cognitive Function in Adolescent Girls in Takalar District, South Sulawesi, Indonesia: Protocol Study

#### **ABSTRACT**

**Background:**Failure to achieve optimal nutritional status in adolescent girls negatively impacts quality of future human resources. National program of Iron-Folic Acid (IFA) tablet supplementation has not shown optimal results due to low compliance and side effects. As an alternative, a food-based supplementation using locally sourced *Moringa oleifera* enriched with royal jelly (MRJ) has been developed. The MRJ formulation is rich in nutrients and has the potential to improve nutritional status and cognitive function. This study evaluates the effect of MRJ on nutritional status and supplement cognitive function in adolescent girls.

**Methods:**This double-blind, randomized controlled trial was conducted among 372 adolescent girls aged 10–19 years from junior and senior high schools in Galesong Selatan, Takalar District, South Sulawesi. Participants were randomly assigned to either the intervention group receiving MRJ capsules (each containing 490 mg*Moringa oleifera*extract and 10 mg*royal jelly*, taken twice per week for 12 months), or the control group receiving weekly IFA tablets (60 mg elemental iron and 400 μg folic acid) following national guidelines. Both groups received standardized nutrition education via TikTok videos. Data collected at baseline, 6 months, and 12 months included anthropometric indicators (BMI-for-age, height-for-age, MUAC), hemoglobin levels (measured using Hemocue), dietary intake (24-hour recall and FFQ), and cognitive function (assessed using the Culture Fair Intelligence Test/CFIT). Adherence was monitored through weekly control sheets verified by teachers, and digital documentation via WhatsApp.

**Discussion:**The study was designed to assess whether MRJ offers a superior, culturally acceptable supplementation strategy compared to IFA. Results will inform local policy and broader applications of food-based interventions to improve adolescent nutrition and cognitive development.

#### **Keywords**

Anemia, Moringa oleifera, Royal jelly, Nutritional status, Cognitive function.

#### **INTRODUCTION**

#### **Background and rationale**

Adolescence is a crucial time characterized by substantial cognitive and psychological development as well as rapid physical growth (1). For these processes to be supported, optimal nutrition is crucial during this phase (2). Long-term health effects of nutritional deficiencies include stunted growth, anemia, and impaired cognitive function, especially in adolescent girls (3.4). Adolescents around the world, particularly girls, face starting nutritional challenges (5). The World Health Organization notes that iron deficiency is the primary cause of anemia in about 30% of teenage girls, a statistic that emphasizes the necessity of focused interventions (6). Adolescent girls in Indonesia continue to suffer from a startingly high rate of chronic energy deficiency (CED); national surveys show that more than 21% of them consume insufficient amounts of energy, which results in less-than-ideal growth and development (7.8).

Long-term nutritional deprivation can result in stunting, which is still a serious problem (9). According to recent studies conducted in Indonesia, among teenage girls between the ages of 16 and 18, the prevalence of stunting can reach 26.9% (10). In addition to limiting physical potential, stunted growth has significant effects on cognitive development, academic achievement, and future economic productivity (11,12). A second chance to lessen the long-term effects of stunting is to address it during adolescence (13). These difficulties are aggravated by anemia, which is primarily brought on by iron deficiency (14). Although the prevalence of anemia among teenage girls in Indonesia declined marginally from 32% in 2018 to 24.1% in 2023, it is still a public health issue (15). Anemia impairs physical activity, cognitive function, and general quality of life by affecting the blood's ability to carry oxygen (16,17). Pregnant girls who have anemia are more likely to experience problems for both the mother and the unborn child (18).

Implementing traditional supplementation programs, such as giving out iron-folic acid tablets, has proven difficult (19). One major obstacle has been low compliance brought on by side effects like gastrointestinal distress (20). Program success is further hampered by poor awareness of the significance of supplementation and restricted access to healthcare facilities (21,22). There is an urgent need for alternative strategies that are both successful and acceptable in the culture (23). A plant that is indigenous to tropical and subtropical areas, Moringa oleifera, has gained attention as a possible remedy (24). Often referred to as "the miracle tree," Moringa is high in antioxidants, vitamins, and iron (25). Research has indicated that it is effective in lowering oxidative stress and

raising hemoglobin levels, both of which improve cognitive function (26,27). The supplement is even more effective when mixed with royal jelly, a nutrient-dense secretion made by honeybees (28). Vitamins B5 and B6 as well as proteins and essential fatty acids, which are found in royal jelly, are known to improve energy metabolism and cognitive function (29).

Adolescent nutrition programs can take a new approach by incorporating Moringa Oleifera Enriched Royal Jelly (MRJ) (30). Because of its natural origins and ease of consumption, MRJ is less likely to cause side effects than traditional supplements and may be more acceptable to teenagers (27). Furthermore, it has been demonstrated that MRJ promotes neurocognitive development by offering vital nutrients needed for brain function and neurotransmitter synthesis (26,29). Adolescent girls' nutritional needs must be met for both their immediate health and the benefit of society as a whole (3.12). Their nutritional status as expectant mothers has a direct effect on the development and health of the offspring (18,22). Improving adolescent girls' nutritional status helps end the intergenerational cycle of malnutrition, which boosts economic growth and human capital (13,30). The purpose of this study is to assess how MRJ supplementation affects the nutritional status and cognitive function of teenage girls in Galesong Selatan, Takalar Regency.

#### **Objectives**

The general objective of this study is to assess the effectiveness of Moringa Oleifera Enriched Royal Jelly (MRJ) supplementation in improving the nutritional status, hemoglobin (Hb) levels, and cognitive function of adolescent girls in Takalar District, South Sulawesi, Indonesia. The study aims to evaluate whether MRJ supplementation, when administered over a 12-month period, can lead to significant improvements in these critical health and cognitive outcomes.

#### **Study Design**

This study employs a true experimental design with a randomized controlled double-blind pretest-posttest approach. Baseline data collection was conducted in the first year, followed by a 12-month intervention during the second and third years. Participants were randomly assigned to two groups: the intervention group received Moringa Oleifera enriched Royal Jelly (MRJ) capsules (containing 500 mg of moringa leaf extract and 10 mg of royal jelly, 2 capsules per week), while the control group received iron-folic acid (IFA) tablets at a dose of 500 mg per week. Both groups received standardized nutrition education through TikTok videos. The intervention was conducted

in a double-blind manner using coded packaging. Nutritional status was evaluated at month 6, and comprehensive assessments of nutritional status and cognitive function were conducted before and after the 12-month intervention.

#### **METHODS: PARTICIPATION, INTERVENTIONS, AND OUTCOMES**

#### Study setting

The study was conducted in Galesong Selatan, Takalar Regency, from July to November 2024, involving two schools: SMAN 13 Takalar and SMPN 3 Galesong Selatan. These schools were chosen due to their representativeness of the adolescent population in both urban and semi-urban settings. Ethical considerations ensured confidentiality regarding specific school identification.

#### **Eligibility Criteria**

Sampling in this study was conducted using purposive sampling technique. After determining the study location, nurses were selected purposively. To be eligible for the study, participants must meet the following criteria:

- (1) Age 10-19 years
- (2) Adolescent girls' who are active in grades 1 and 2 (junior high and senior high)
- (3) Severe nutritional or health conditions (eg, severe anemia, severe malnutrition, allergies), determined through clinical history and validated self-reports.

#### Who will take informed consent?

The researcher and/or enumerator will obtain informed consent from adolescent girls who fit the criteria. Each student's willingness is included in their informed consent, which has been approved by their parents and teachers (class advisors). Following clear explanations of the purpose of the study and the procedure, both the participants and their guardians are given.

## Additional consent provisions for collection and use of participant data and biological specimens

The study was conducted with the knowledge and permission of relevant authorities, including the Takalar District Education Office for junior high schools, the Provincial Education Office for senior high schools, and Bontokassi Primary Health Center, as the selected schools falling under its jurisdiction.

Approval was also obtained from each participating school. Participants' data and biological specimens were anonymized and securely stored. Additional explicit consent was provided

obtained for the use of biological specimens in further analyses, ensuring transparency and compliance with ethical standards.

#### Interventions

#### **Explanation for choice of comparators**

Indonesia's national program on nutritional supplementation includes the "Aksi Bergizi" initiative, which provides iron supplementation through the distribution of Iron-Folic Acid (IFA) tablets to adolescent girls. This intervention aims to increase hemoglobin levels and prevent anemia. IFA tablets are distributed regularly under the supervision of school health personnel to ensure compliance (97). Adolescent girls are required to report their intake, and health staff provide counseling in case of problems or complaints. In addition to distribution, the program offers education on the importance of iron supplementation. Adolescents receive explanations on how the IFA tablets work, their benefits, and ways to manage possible side effects (98).

The Iron-Folic Acid Supplementation Program for adolescent girls is a crucial effort to prevent and address anemia. Anemia among adolescent girls remains a serious public health concern, especially in developing countries like Indonesia. This condition can lead to adverse outcomes such as reduced concentration, lower academic performance, and other health issues. Therefore, IFA supplementation serves as a vital preventive strategy (99).

The supplementation involves providing tablets containing iron and folic acid to adolescent girls on a regular basis. The dosage depends on whether the purpose is prevention or treatment. For prevention, which targets adolescent girls without anemia, the tablets typically contain 60 mg of elemental iron and 400 mcg of folic acid, taken once weekly for one year. This dosage is designed to meet daily nutritional needs and prevent iron deficiency during periods of rapid growth (100). For treatment, adolescent girls diagnosed with anemia receive a higher dose—generally 60 mg of elemental iron and 400 mcg of folic acid taken daily for three months, or as advised by healthcare providers. The therapeutic goal is to rapidly raise hemoglobin levels and address existing anemia (101).

The distribution process begins at the local health office, where IFA tablets are delivered to schools through community health centers or other healthcare facilities. Upon arrival at the school, health personnel are responsible for distributing the tablets to registered adolescent girls. An orientation program is provided to students and parents at the beginning, explaining the importance of IFA

supplementation, proper intake methods, and the associated health benefits. This is intended to ensure that all stakeholders understand the program's purposes and procedures (102).

Although the program has demonstrated effectiveness in several studies when implemented according to guidelines, challenges remain in practice. Unequal distribution of IFA tablets has resulted in limited access for some adolescent girls. Low compliance, driven by limited knowledge, aversion to the tablets, and side effects, have also significantly hindered the success of the program.

#### Intervention description

#### The study will involve two groups:

- 1.**Control Group**: Participants will follow the *Nutritious Action* program, which includes Iron-Folic Acid (IFA) supplementation and video-based education using the TikTok application.
- 2.**Intervention Group**: Participants will follow the *Nutritious Action* program, but IFA supplementation will be substituted with MRJ (Moringa-Royal Jelly). They will also receive video-based education via TikTok, using the same content as the control group.

The IFA tablet contains 60 mg of elemental iron and 400 µg of folic acid. Meanwhile, MRJ (500 mg) consists of 490 mg Moringa extract and 10 mg Royal Jelly extract, and contains various nutrients such as iron (9.72 mg), vitamin C (46.2 mg), zinc, calcium, flavonoids, polyphenols, antioxidants, beta-carotene, and other essential vitamins and minerals.

#### Criteria for discontinuing or modifying allocated interventions

Adolescent girls enrolled in the clinical trial who experience allergic reactions or adverse effects reported in either study group will be referred to a midwife or physician for evaluation and guidance on whether to continue participation or withdraw from the study. Participants are free to withdraw at any time and for any reason without any consequences.

#### Strategies to control interventions

Schools and students for both the intervention group (MRJ) and the control group (IFA) will be selected to participate in the study. One teacher from each school—preferably the School Health

Unit (SHU) teacher—will be invited to assist and supervise students consuming the supplements at school on a designated day each week.

Each student will receive two capsules per week—one to be consumed at school under supervision, and one to be taken home as a backup in case the student is absent on the scheduled supplement day the following week.

Each participant will be provided with a monitoring sheet, which will be signed by the supervising teacher if the supplement is consumed at school. If consumed at home, the student is required to submit photographic documentation with a real-time timestamp. This documentation will be reviewed by the supervising teacher and acknowledged with a signature on the student's compliance sheet.

If a student is absent on the scheduled day, he may take the supplement at home with appropriate documentation, which will be verified by the teacher for validation and recorded on the control sheet.

A WhatsApp (WA) group will be created for each study group. Through these groups, the researcher will send regular reminders to students to take their capsules on the designated day. In addition, educational links related to anemia in adolescent girls—including its impacts, prevention, and the benefits of the given supplements—will be shared monthly. A total of 12 different educational videos will be sent throughout the study period.

Biweekly school visits will be conducted to evaluate implementation, confirm supplement consumption, and identify any barriers or difficulties encountered by students in taking the capsules.

#### **Operational Definition**

- a) Moringa Extract Enriched Royal Jelly (MRJ) Administration
  - The intervention group will receive a capsule formulation (500 mg) containing 490 mg of *Moringa oleifera*extract and 10 mg of royal jelly extract. Each capsule contains essential nutrients such as iron (9.72 mg), vitamin C (46.2 mg), zinc, calcium, flavonoids, polyphenols, antioxidants, beta-carotene, and other vitamins and minerals. The capsules will be administered to anemic adolescent girls at a dosage of two capsules per week over a 12-month period.
- b) Iron and Folic Acid (IFA) Administration

IFA tablets (containing 60 mg of elemental iron and 400  $\mu$ g of folic acid) will be distributed to adolescent girls according to the national program. Both MRJ and IFA will be administered under a double-blind design, ensuring that both supplements appear visually identical in capsule form.

#### c) Compliance Monitoring

To assess adherence, a consumption control sheet will be provided to each participant by the researcher or enumerator. This sheet will be checked and signed by the assigned supervising teacher. If capsules are consumed at school, the teacher will sign the sheet. If taken at home, the participant must document the intake with a time-stamped photo, which the teacher will verify and sign accordingly.

#### d) Nutrient Intake

Nutrient intake refers to the total consumption of macronutrients (energy, carbohydrates, fats, and proteins) by adolescent girls in a day. This will be measured using a 24-hour dietary recall and a Food Frequency Questionnaire (FFQ), and compared with the recommended dietary allowance (RDA) for their age.

#### e) Nutritional Status

Includes Body Mass Index-for-Age (BMI/A), Height-for-Age (H/A), Mid-Upper Arm Circumference (MUAC), and hemoglobin levels:

- Body weight will be measured using a SECA digital scale.
- Height will be measured with a stadiometer.
- MUAC will be assessed using a standard MUAC tape.
- Hemoglobin levels (Hb) will be measured using a Hemocue device by trained enumerators.

#### f) Cognitive Function

Cognitive function will be assessed using the standardized *Culture Fair Intelligence Test* (CFIT) questionnaire. The test will be administered and analyzed directly by a licensed psychologist from Hasanuddin University.

#### **Study Subjects**

The population in this study includes all female students at junior high schools (SMP) and senior high schools (SMA) in Galesong Selatan Subdistrict, Takalar Regency, South Sulawesi

Province. The sample size in this study is calculated using the formula for estimating the mean difference between two paired groups, as proposed by Lemeshow and Wanga (1991), as follows:

n = 
$$\frac{\sigma^{2}(z_{1-\infty/2} + z_{1-\beta})^{2}}{(\mu_{0} - \mu_{1})^{2}}$$
=2 x \frac{1.23^{2}(1.9 + 0.9)^{2}}{(11.42 - 10.85)^{2}}
=\frac{3.02(7.84)}{(0.57)^{2}}
=\frac{23.7}{0.33}
=71.8 = 72

Note:

n : Sample Size

Ó : Standard deviation 1.23

Z1-α: Significance level 95%(1.96) Z1-

 $\beta$ : Power of the test 90%(0.9)  $\mu$ 1

: Mean hemoglobin level in the MRJ intervention group (11.42 g/dl) :

 $\mu$  2 Mean hemoglobin level in the placebo intervention group (10.85 g/dL)

The sample size calculation was based on the standard deviation and mean values from previous studies for the dependent variable. Based on this calculation, the required number of participants was 72. However, to anticipate potential dropouts (DO), a 10% increase (7 participants) was added, resulting in a total of 79 participants. Therefore, each group will consist of 79 samples: 79 participants in the intervention group and 79 in the control group.

This study will collect two types of data: primary and secondary data. Primary data will be obtained through questionnaires distributed to the respondents and analyzed using SPSS version 26. Secondary data will be collected from relevant literature or previous research studies. The study will be conducted in three phases:

1) Preparation and Baseline Data Collection

This stage involves assigning students to the intervention and control groups. Baseline data collection will be conducted at the selected schools for each group, including

measurements of nutritional status (body weight, height, dietary intake, and hemoglobin levels) and cognitive function levels.

#### 2) Intervention Phase and Mid-Evaluation

This phase involves interventions for the two groups: the intervention group receiving MRJ and the control group receiving IFA (iron and folic acid tablets). The MRJ and IFA capsules will be provided in pre-packaged bottles containing 10 capsules, to be consumed over 5 weeks. New supplies will be distributed every 5 weeks up to the 48th week (12 months).

#### 3) Extended Intervention and Final Evaluation Phase

After 12 months, the nutritional and cognitive status of the adolescent girls will be reevaluated. This will allow assessment of improvements at 6-month intervals and determination of the most effective supplementation duration.

#### **Instruments and Intervention Materials**

Materials used in this study were MRJ and IFA capsules purchased as finished products. IFA contains 200 mg ferrous sulfate (equal to 60 mg elemental iron) and 0.25 mg folic acid. MRJ contains 500 mg moringa and 10 mg royal jelly. Both were packed in identical capsules in terms of shape, color, and size to ensure blinding, so no visual difference between them. Capsules were supplied by trusted manufacturer and randomly coded by independent third party to maintain confidentiality during intervention. Before distribution, materials were tested for quality to ensure safety and formulation consistency.

Instruments used included Kobo questionnaire, 24-hour recall and FFQ, anthropometric tools: digital scale (Seca) for weight, stadiometer for height, MUAC tape, Hemocue for hemoglobin levels, CFIT for cognitive test, and checklist sheets for monitoring MRJ and IFA capsule consumption compliance.

#### **Nutrition and Anemia Education**

Balanced nutrition and anemia education will be conducted both offline and online. Offline education will be given before and after the intervention (pre-posttest) through a 30–45-minute lecture. Each session will include ice-breaking and a quiz with prizes to make the learning process interactive and enjoyable. Online education will run throughout the 12-month intervention via TikTok-based educational video links. These links will be shared with

study subjects through a WhatsApp group. Video updates will be sent every two weeks. The education topics, both offline and online, will remain the same, including:

#### **Topic 1: Balanced Nutrition**

Optimal nutrient intake is essential for the body's growth and development. Dietary patterns should focus on consuming a balanced diet—daily meals that contain nutrients in types and amounts that meet the body's needs.

#### **Four Pillars of Balanced Nutrition:**

- 1. Consume a variety of foods.
- 2. Practicing clean and hygienic living.
- 3. Engaging in physical activity.
- 4. Monitor body weight regularly.

#### **Topic 2: My Plate Contents**

A guide to food diversity and recommended portion sizes for each meal. Each plate should consist of 2/3 staple foods and vegetables, and 1/3 side dishes and fruits. It's also important to limit sugar, salt, and fat intake and drink adequate water.

#### **Topic 3: Protein: The Body Builder**

Protein is necessary for the formation of new cells, cell maintenance, and boosting immunity.

Protein sources include animal proteins such as meat, fish, and eggs, as well as plant-based proteins such as tofu, tempeh, and legumes. A balanced intake of both animal and plant proteins is recommended.

#### **Topic 4: Healthy Breakfast**

Breakfast fulfills 20–25% of daily calorie needs. A healthy breakfast includes sources of carbohydrates, proteins, fats, and vitamins/minerals in appropriate portions.

#### **Topic 5: Physical Activity**

Regular physical activity helps maintain fitness, boosts metabolism, and prevents obesity. The WHO recommends 60 minutes of daily physical activity for children and adolescents.

#### Topic 6: Food and Beverage Labels

Food labels help consumers understand nutritional content, monitor sugar, salt, and fat limits, and ensure food safety. Nutrition literacy is crucial for making informed dietary choices.

#### **Topic 7: School Canteens and Healthy Snacks**

Avoid snacks with artificial coloring, reused cooking oil, and excessive sugar, salt, or fat content. Choose snacks from clean and safe vendors.

#### Topic 8: Fruit and Vegetable Consumption

Fruits and vegetables are rich in vitamins, minerals, and fiber. It is recommended to consume 3–4 servings of vegetables and 2–3 servings of fruit daily to maintain health and prevent disease.

#### **Topic 9: Anemia and Iron**

Anemia is often caused by iron deficiency. Prevention can be done by consuming iron-rich foods such as red meat, spinach, and legumes.

#### **Topic 10: Micronutrients**

Vitamins and minerals are essential for bodily functions, even in small amounts. Consume foods rich in micronutrients such as leafy greens, fruits, and legumes.

#### Topic 11: Sugar, Salt, and Fat

Limit intake of sugar (maximum 50 grams/day), salt (5 grams/day), and fat (67 grams/day). Excessive consumption increases the risk of chronic diseases.

#### **Topic 12: Personal Hygiene**

Clean living includes habits such as handwashing, food hygiene, and personal health maintenance. Good hygiene reduces the risk of infection and supports overall health.

#### **Data Analysis**

The primary data collected were then processed through several stages of data handling as follows:

- a. Editing: The results obtained from interviews or questionnaires were first edited. If there were any incomplete data or missing information, corrections were made efficiently. If it was not possible to re-interview the respondent, the questionnaire was excluded from the dataset.
- b. Coding: Each item in the questionnaire was assigned a numeric code to facilitate data processing and analysis.
- c. Tabulation: The data were grouped and presented in tabular form in accordance with the research objectives, making it easier to analyze.

- d. Processing: In this stage, the responses from participants, which had been translated into numerical form, were processed for analysis.
- e. Cleaning: The data entered into the master table were rechecked, including verification of data entries and codes, to minimize errors during the data input process. If incorrect coding was found, it was corrected or removed based on the original questionnaire.

After the data processing phase, data analysis was conducted using SPSS, employing univariate, bivariate, and multivariate analyses.

- Univariate analysis aims to obtain an overview and describe the characteristics of
  each research variable, including age, education, income, occupation, parity,
  pregnancy history, dietary intake, mid-upper arm circumference, gestational age,
  infant length, and birth weight. This analysis generated frequency distribution tables
  and percentages for each variable.
- Bivariate analysis was conducted to assess the differences in means before and after
  the intervention within each group. A paired t-test was used if the data were
  normally distributed, while the Wilcoxon test was used for non-normally distributed
  data. For categorical data, the McNemar test was applied. To compare the mean
  changes between the three groups, One Way ANOVA was used for normally
  distributed data, and the Kruskal-Wallis test for non-normally distributed data.
- Multivariate analysis was performed to examine the effect of independent variables on the dependent variable using Logistic Regression analysis.

#### **Quality Control**

Quality control is directed toward minimizing errors that may arise from sampling factors (sampling error) or alpha errors, which include errors due to an inadequate sample size or an unrepresentative sample that does not accurately reflect the population. In addition, quality control also aims to address systematic errors or beta errors, which may originate from the measuring instruments, the measurer, or the object being measured.

Standardization of the instruments used was conducted through validity testing on adolescent girls. Prior to the implementation of the research, the researcher submitted formal requests and obtained approval from the relevant authorities, including the local health office,

schools, and community health centers (Puskesmas). Once permission was granted, an informed consent form was provided and signed by each respondent as a confirmation of their voluntary participation.

#### **Research Ethics**

This study was conducted after obtaining ethical clearance from the Health Research Ethics Committee of the Faculty of Public Health, Hasanuddin University, with Ethical Approval Number 2739/UN4.14.1/TP.01.02/2024, dated September 30, 2024.

#### **Research Flow Chart**



Participants in the intervention group were included in the *Nutritious Action* activities, which also incorporated educational sessions. During each scheduled group meal (as per prior agreement), each subject received 2 capsules to be taken immediately and an additional 1 capsule to take home for the following week. This third capsule was intended to anticipate possible absence in the subsequent session; if a participant was absent, she was instructed to consume the capsule at home and provide photo documentation as proof, which was then initialed by the teacher on the compliance sheet.

### WhatsApp Group Formation ed as a reminder platform and an educa

WhatsApp groups were created as a reminder platform and an educational channel, through which educational video links were shared regularly with participants.



Figure 1. Research Flow Diagram

#### **Research Timeline**

In the first year, the study begins with field preparation activities, including coordination with schools, healthcare personnel, and enumerators. This was followed by the collection of baseline data to assess the nutritional status and cognitive function of adolescent girls. The collected data were then analyzed during the baseline data analysis phase and used to prepare the initial findings report. The baseline results also served as the foundation for developing journal articles and scientific publications. At the end of the first year, the intervention phase was initiated, accompanied by a monitoring process of capsule consumption by participants.

In the second year, activities commenced with intervention preparation, followed by full implementation of the intervention. A midline evaluation was conducted in the sixth month to assess the preliminary effects of the intervention on dietary intake and nutritional status. The data from this evaluation were analyzed in the six-month intervention data analysis phase and compiled into reports and scientific articles. Publication activities continued, along with the preparation and implementation of the 12-month intervention evaluation toward the end of the second year.

In the third year, the follow-up 12-month evaluation was carried out to assess the final outcomes on dietary intake, nutritional status, and cognitive function of adolescent girls postintervention. The data were analyzed in the 12-month intervention data analysis phase, and the results were compiled into the final report and scientific articles. The final stage of this research involved the dissemination of findings through publications in national and international scientific journals. Outcomes

#### **Participant Characteristics**

The study enrolled 372 participants, with a mean age of 14.5 years (±1.2). Baseline characteristics, including nutritional status, socioeconomic background, and dietary patterns, were comparable between the intervention and control groups.

#### **Nutritional Status**

Participants receiving MRJ supplementation showed significant improvements in weight-for-age and height-for-age Z-scores compared to the control group (p < 0.05). MUAC measurements also indicated better chronic energy deficiency outcomes in the intervention group.

#### **Cognitive Function Scores**

Cognitive function, as assessed by CFIT, improved significantly in the MRJ group compared to the control group.

#### REFERENCES

- 1.Patton GC, Sawyer SM, Santelli JS, et al. Our future: a Lancet commission on adolescent health and wellbeing. Lancet. 2016;387(10036):2423–78.
- 2.World Health Organization. Nutrition in adolescence: issues and challenges for the health sector. Geneva: WHO; 2005.
- 3.Black MM. Micronutrient deficiencies and cognitive functioning. J Nutr. 2003;133(11 Suppl 2):3927S–31S.
- 4.Best C, Neufingerl N, Van Geel L, van den Briel T, Osendarp S. The nutritional status of schoolaged children: why should we care? Food Nutr Bull. 2010;31(3):400–17.
- 5.UNICEF. The State of the World's Children 2019: Children, food and nutrition. New York: UNICEF; 2019.
- 6. World Health Organization. Anaemia in women and children. Geneva: WHO; 2023.
- 7.Health Research and Development Agency. Basic Health Research 2018. Jakarta: Ministry of Health, Republic of Indonesia; 2018.
- 8.Ministry of Health of the Republic of Indonesia. Indonesia Health Profile 2023. Jakarta: MoH: 2024.
- 9.Dewey KG, Begum K. Long-term consequences of stunting in early life. Matern Child Nutr. 2011;7(Suppl 3):5–18.
- 10.Hadju V, Salmah AU, Natsir R, et al. Stunting and its risk factors among adolescent girls in South Sulawesi. Indonesian Community Nutrition Media. 2020;5(2):59–66.
- 11.Walker SP, Chang SM, Powell CA, et al. Effects of early childhood psychosocial stimulation and nutritional therapy on cognition and supplement education in growth-stunted Jamaican children. Lancet. 2005;366(9499):1804–7.
- 12.Grantham-McGregor S, Cheung YB, Cueto S, et al. Developmental potential in the first 5 years for children in developing countries. Lancet. 2007;369(9555):60–70.
- 13.Prentice AM, Ward KA, Goldberg GR, et al. Critical windows for nutritional interventions against stunting. Am J Clin Nutr. 2013;97(5):911–8.
- 14.Stoltzfus RJ. Iron deficiency: global prevalence and consequences. Food Nutr Bull. 2003;24(4 Suppl):S99–103.
- 15.Ministry of Health of the Republic of Indonesia. Indonesia Nutrition Status Survey (SSGI) 2023. Jakarta: MoH; 2024.
- 16.Beard JL. Iron deficiency alters brain development and functioning. J Nutr. 2003;133(5 Suppl 1):14685–72S.
- 17. Haas JD, Brownlie T. Iron deficiency and reduced work capacity: a critical review of the research to determine a causal relationship. J Nutr. 2001;131(2S-2):676S–88S.
- 18.Allen LH. Anemia and iron deficiency: effects on pregnancy outcome. Am J Clin Nutr. 2000;71(5 Suppl):1280S–4S.
- 19.Bhan MK, Sommerfelt H, Strand T. Micronutrient deficiency in children. BMJ. 2001;323(7308):1408–12.
- 20.Ridwan E, Madanijah S, Briawan D, Dwiriani CM. Effect of Fe supplementation on Hb levels and adherence to Fe tablet consumption in adolescent girls. Indonesian Nutrition. 2014;37(2):125–34.
- 21.Titaley CR, Dibley MJ, Roberts CL, Hall J, Agho K. Iron and folic acid supplements and reduced early neonatal deaths in Indonesia. Bull World Health Organs. 2010;88(7):500–8.

- 22.Kurniawan Y, Briawan D, Madanijah S. Role of family support in adherence to iron tablet consumption. J Nutrition and Food. 2016;11(2):105–12.
- 23. Nurbaya S, Yusuf SM, Hadju V, et al. Cultural acceptability and compliance of adolescent iron supplementation in South Sulawesi. J Nutr College. 2020;9(1):1–8.
- 24. Saini RK, Sivanesan I, Keum YS. Phytochemicals of Moringa oleifera: a review of their nutritional, therapeutic and industrial significance. 3 Biotech. 2016;6(2):203.
- 25.Gopalakrishnan L, Doriya K, Kumar DS. Moringa oleifera: a review on nutritional importance and its medicinal applications. Food Sci Hum Wellness. 2016;5(2):49–56.
- 26.AR's son, Hadju V, Santoso LA. The effect of Moringa leaf powder supplementation on hemoglobin levels in adolescent girls. Indian J Public Health Res Dev. 2019;10(8):2805–8.
- 27.Faizal A, Mutalib AR, Hamzah Z, et al. Combination of royal jelly and moringa improves hemoglobin levels and reduces oxidative stress in anemic rats. J Appl Pharm Sci. 2022;12(1):74–80.
- 28.Ramadan MF, Al-Ghamdi A. Bioactive compounds and health-promoting properties of royal jelly: a review. J Funct Foods. 2012;4(1):39–52.
- 29.Ahmad S, Campos MG, Fratini F, et al. New insights into the biological and pharmaceutical properties of royal jelly. Int J Mol Sci. 2020;21(2):382.
- 30.Yusuf S, Hadju V, Arsyad DS, et al. Integrating MRJ (Moringa + Royal Jelly) supplementation in school-based nutrition programs: feasibility and early outcomes. J Nutr Educ Behav. 2024;56(1):e45–e52.
- 31.Lemeshow S, Wanga DW. Adequacy of sample size in health studies. Chichester: John Wiley & Sons; 1991.

#### QUESTIONNAIRE

#### RESEARCH RESPONDENT CONSENT SHEET

The undersigned below:

"The Effect of Giving Moringa Oleifera Enriched with Royal Jelly on the Nutritional Status and Cognitive Level of Adolescent Girls"

| Name | | : | | | |
|---|---|---|---|---|---|
| Age | | : | | | |
| Phone number | | : | | | |
| Address | : | | | | |
| this research. Th<br>months.<br>After receiving t | nis explanation includes<br>he explanation, I hereb | the objectives, benefits | oportunity to ask questions, and effects of this rese<br>this study and am willing<br>this study and am willing | arch. This research proc<br>og to follow the blood sa | edure will take 12<br>mpling procedure, |
| Thus I make this | s statement in truth. | | | | |
| | | | | Takalar | 2024 |
| Res | spondents/ Students | | | | |
| (. | ) | | | | |



#### QUESTIONNAIRE FOR NUTRITIONAL INTERVENTION RESEARCH FOR ADOLESCENT GIRLS ANEMIA

#### In Takalar Regency in 2024

| | | BLOCK I. DATA COLLECTOR DESCRIPTION | | |
|---|---|---|---|---|
| 1 | Data collection date | | | 00-00-000 |
| 2 | Name | | | |
| 3 | Mobile phone number | | | |
| | | BLOCK II. CHARACTERISTICS OF SUBJECTS AND PAR | ENTS | |
| 1 | Name | | | |
| 2 | Date of birth | | | 00-00-000 |
| 3 | Age | | | |
| 4 | School name | | | |
| 5 | Class (school) | | | |
| 6 | Home address | | | |
| 7 | Phone number | | | |
| 8 | Number of Family Members Living at | Home | | |
| 9 | What order do you come in your family | | | |
| 10 | How many brothers and sisters do you have | | | |
| | Fathe | r | | Mother |
| 11 | Name | | | |
| 12 | Mobile phone number | | | |
| 13 | Date of birth | 30-000 | | 00-00-000 |
| 14 | Father's Education | | | |
| 15 | Mother's Education | | | |
| | Education Options No/Not YetAt School Not graduated from elementary school/Islamic elementary school Graduated from Elementary School/Islamic Elementary School Graduated from junior high school/Islamic junior high school Graduated from high school/Islamic high school GraduatedDI,DII,DIII GraduateDIV/PT | Job Options 1.Doesn't work 2. School 3.Civil Servants/TNI/Polri/BUNM/BUMD 4. Private employees 5.Self-employed 6. Farmer/ Farm Worker 7.Fisherman 8.Laborer/Driver/Motorbike Taxi/Maid | Family Income Op<br>0 - Rp. 500,000.00<br>2. > Rp. 500,000.00 -<br>3. > Rp. 1,000,000.00<br>4. > Rp 2,000,000.00<br>5. > Rp. 3,000,000.00<br>6. ≥ Rp 4,000,000.001 | Rp. 1,000,000.00<br>- Rp. 2,000,000.00<br>- Rp 3,000,000.00<br>- Rp. 4,000,000.00 |
| 16 | Father's occupation | | | |
| 17 | Mother's Job | | | |

| 18 | How Much is the Family Income? | |
|---|---|---|
| 19 | What is the main type of water source for all your household needs? (mark one option): | |
| | a. Tap water/PDAM f. Protected springs b. Retail tap water/purchased g. Unprotected springs c. Boreholes/pumps<br>h. Rainwater storage d. Protected dug wells i. River/lake/irrigation water | |
| 20 | How is the use of household defecation facilities? | |
| | a. Owned by yourself d. Shared with a neighbor b. Shared with others e. None | |
| 21 | How many times does the family provide food in a day? | |
| | BLOCK III. PMS Status of Adolescent Girls | |
| 1 | Have you menstruated yet? 1 = Yes, 2 = Not yet | |
| 2 | When did you first have your period? (dd-mm-yr) | |
| 3 | How long is menstruation? | |
| 4 | Complaints 1-2 weeks before menstruation (1 = Yes, 2 = No) | |
| 5 | Menstrual complaints (1 = Yes, 2 = No) | |
| 6 | Mother/sister experiences complaints during menstruation | |
| PMS Sy | mptom Scale | |
| 1 = No | t experienced, Scale 2 = Very light, Scale 3 = Light, Scale 4 = Moderate, Scale 5 = Severe, Scale | 6 = Extreme |
| 1 | Breasts feel sore, tense, enlarged or swollen | |
| 2 | Feeling unable to adjust or overwhelmed in daily activities | |
| 3 | Feeling stressed | |
| 4 | Easily offended or easily angered | |
| 5 | Feeling sad or disappointed | |
| 6 | Back pain, aches or stiffness in the joints | |
| 7 | Weight gain | |
| 8 | Stomach feels sore or uncomfortable | |
| 9 | Swelling in certain areas of the body | |
| 10 | Feeling bloated | |
| | BLOCK IV. Signature Compliance Questionnaire | |
| 1 | Have you ever received a signature? | 1 YES, 2 NO |
| 2 | Do you currently have a signature? | 1 YES, 2 NO |
| 3 | Since when did you get your signature? | |
| 4 | How many signatures were obtained? | 1 tablet/week |
| | | monthly table |
| 5 | Have you ever taken TTD? | 1 YES, 2 NO |
| 6 | Are you currently taking TTD? | 1 YES, 2 NO |
| 7 | When do you take TTD? | Once a week |
| | | Once every 10 days |
| | | very |

| 8 | How long have you been taking TTD? | Sunday | |
|---|---|---|---|
| 9 | How much TTD do you consume? | | 1 tablet/week |
| | | | 4 tablets/month |
| 10 | Reasons for Consuming: | | |
| 11 | Reasons Not to Consume: | | |
| 12 | complaints when taking TTD | | |
| | BLOCK V. Nutritional Status of | Adolescent Girls | |
| | Examination Date I | | |
| 1 | Hb | | g/dl |
| 2 | Height | | |
| 3 | close body | | |
| 4 | iLA | | |
| | Block VI Eating P | atterns | |
| | 1= Yes (always done 5- | 7 times/week) | |
| | 2= Sometimes (3-4 t | imes/week) | |
| | 3= Rarely (times | s/week) | |
| | 0= Never | | |
| 1 | According to you, what is meant by breakfast? | . Correct | |
| | Answer: | . Wrong | |
| | <b>Answer:</b> Breakfast is a meal eaten in the morning before starting activities. | | |
| 2 | How often did you eat breakfast in the last week? | the | |
| | | reason | |
| 3 | Does your family usually provide breakfast at home? | the | |
| | | reason | |
| 4 | When you don't have time for breakfast, you bring your own food or do | on't buy snacks at school | |
| 5 | Do you like to snack? | | |
| 6 | How many times do you snack in a day? | | |
| 7 | What time of food do you must often out as a small? | 1. Fried food | |
| / | What type of food do you most often eat as a snack? | 2. Chiki | |
| | | 3. Chocolate | |
| | | 4. Meatballs<br><b>5. Wafe</b> r | |
| | | 6. Biscuits | |

| | | Etc., please mention | |
|---|---|---|---|
| 8 | What are 3 types of food you like? | | |
| | Block VII Physical Activity | y (IPAC) | |
| Answer e<br>are at wo | owing questions will ask you about the time you spent be<br>each question even if you do not consider yourself an ac<br>ork, as part of housework and yard work, traveling from<br>or sports. | tive person. Think abo | out activities you do while you |
| 1 | During the last 7 days, on how many days did you do he activity? such as lifting heavy objects, climbing stairs, and mandato school hours (volleyball, fast cycling, digging and so on) | | days of the week |
| 2 | How much time do you usually spend each day doing vi<br>activity as part of your study activities? | gorous physical | hours / days<br>minutes / day |
| a little h | What kind of strenuous activities do you do? 1. Lifting heavy loads 2. Aerobics 3. Fast cycling 4. others please specify bout the moderate physical activity you did in the last 7 carder than usual. For example, carrying a light load, cyclite physical activity makes you breathe a little harder than | ling or playing sports. | |
| do it for | at least 10 minutes. | | |
| 4 | During the past 7 days, on how many days did you do modera such as carrying light loads, cycling regularly, or playing doublinclude walking. | | days of the week |
| 5 | How much time do you usually spend doing moderate រុ<br>a day? | ohysical activity | hours / days<br>minutes / day |
| 6 | What kind of moderate activities do you do? 1. Carrying light loads 2. Leisurely cycling 3. Mopping 4. Washing 5. Others, please specify | | |
| 7 | During the last 7 days, on how many days did you walk for minutes at a time? | at least 10 | days of the week |
| 8 | How much time do you usually spend walking in a day? | | hours / days<br>minutes / day |
| 9 | How much time do you usually spend sitting on weekda | ays? | hours / days<br>minutes / day |

| 10 | What kind of light activities do | you do? | | |
|---|---|---|---|---|
| | 1. Sweeping | | | |
| | 2. Walking | | | |
| | 3. Others, please specify | | | |
| | | Block VIII Food Believe and Food Taboo | | |
| 1 | Are there certain types of food tha | t you are prohibited from consuming? | | |
| | . Yes | | | |
| | . No | | | |
| 2 | What foods are you not allowe | ed to eat? | | |
| | weld: | | | |
| 3 | Are there any special foods that | 1. Yes, please specify | | _ |
| | you consume at certain times<br>(celebratory holidays/religious | 2. No<br>Reason : | | |
| | events/during menstruation, etc.) | (ed5011 . | | |
| | | | _ | |
| 4 | Where did you get the | | | |
| 4 | Where did you get the information about consuming | <ol> <li>Mother</li> <li>Other family (father, brother, grandmother, etc.)</li> </ol> | | |
| | what is that special food? | 3. Neighbors | | |
| | | <ul><li>4. Peers</li><li>5. Others, please specify</li></ul> | | |
| 5 | What are the 5 types of food that you often o | | | |
| | | Block IX PSP Teen Girls | | |
| Knowle | edge (1= YES, 2= NO) | | | |
| 1 | dress neatly and cut nails <i>No</i> on | e of the healthy and clean living habits | | |
| 2 | It is recommended that we drink 5 glasses of | water every day | | |
| 3 | Breakfast is needed as the main | source of energy before starting daily activitie | 25. | |
| 4 | Indonesia has a balanced nutrition gu | ideline consisting of four pillars of balanced nutriti | on, namely: consuming | |
| | 7 | ysical activity, clean living habits, and monitorin | g body weight. | |
| 5 | Teenagers who don't like vegetables tend to be fat as adults | | | |
| 6 | It is recommended to do physical activity or exercise at least once a week for 1 hour. | | | |
| 7 | We don't need to limit our consumption of sugar, salt and fat because they are beneficial for our bodies. | | | |
| 8 | anemia is a condition with hem | oglobin levels lower than normal values | | |
| 9 | anemia/insufficient blood is ca | used by not eating enough foods rich in iro | n | |
| 10 | you and the symptoms of anemia that you see ar | e fatigue, exhaustion, lethargy, inattention and weakness | | |

| 11 | Anemia in adolescents can have an impact on the ability to concentrate. |
|---|---|
| 12 | Teenagers experience menstruation so they need to be given additional iron (TTD) |
| 13 | The correct way to wash your hands is to use running water and soap |
| 14 | Lack of nutrition in adolescent girls can lead to malnutrition during pregnancy. |
| 15 | If the environment is dirty and unhygienic, a person can easily catch a disease. |
| Attitude | e (1= AGREE, 2= DISAGREE) |
| 1 | Dressing neatly and cutting nails has no effect on my health. |
| 2 | Drinking 5 glasses of water is enough to meet my needs |
| 3 | Breakfast is important to me, because otherwise I will have difficulty concentrating at school. |
| 4 | You don't need to worry if someone is tired, weak, lethargic and pale. |
| 5 | I have to eat vegetables every day to improve my digestion |
| 6 | I don't consider the nutritional and health information on food labels when choosing food. |
| 7 | I will choose foods with less sugar, salt and fat, even though they are not as delicious as foods high in sugar, salt and fat |
| 8 | I can apply the 4 pillars of balanced nutrition guidelines in everyday life. |
| 9 | The balanced nutrition pyramid helps me choose the right foods |
| 10 | Eating tofu and tempeh alone is enough to build cells and tissues in our bodies. |
| 11 | I need to eat vegetables and fruit to avoid constipation |
| 12 | If your hands don't look dirty, washing them with running water is enough. |
| 13 | Now I don't have to worry about my nutritional status as a future parent. |
| 14 | I need to pay attention to the cleanliness of the surrounding environment because it will affect my health. |
| 15 | I don't consider the nutritional and health information on food labels when choosing food. |
| Practic | e: a= Always, b= Often, c= Sometimes, d= Rarely, e= Never |
| 1 | How often do you dress neatly and cleanly? |
| 2 | How often do you drink 8 glasses of water per day? |
| 3 | How often do you eat breakfast before 9 am? |
| 4 | How often do you consume sources of iron (red meat, chicken liver, iron tablets)? |
| 5 | How often do you eat vegetables? |
| 6 | Do you read food labels before deciding to buy packaged food? |
| 7 | How often do you drink sugary drinks? |
| 8 | How often do you weigh yourself? |
| 9 | How often do you use the balanced food pyramid as a food guide? |
| 10 | How often do you consume animal protein sources? (eggs, red meat, chicken) |
| 11 | How often do you do continuous physical activity for at least 30 minutes? |
| 12 | How often do you eat fruit? |
| 13 | Do you wash your hands after using the bathroom? |
| 13 | Do you wash your hands after using the pathroom? |

| 14 | How often do you search for nutrition and health information? |
|---|---|
| 15 | Do you help clean up your environment? |
| | Block X Self Efficacy of Adolescent Girls |
| | (1= SURE, 2= NOT SURE) |
| 1 | How confident are you that you can dress neatly and cleanly every day? |
| 2 | How confident are you in drinking 8 glasses of water per day? |
| 3 | How confident are you in having breakfast before 9 o'clock? |
| 4 | How confident are you in consuming sources of iron at every meal (red meat, chicken liver, iron tablets)? |
| 5 | How confident are you in eating vegetables at every meal? |
| 6 | How confident are you in reading food labels before deciding to buy packaged food? |
| 7 | How confident are you about weighing yourself once a month? |
| 8 | How confident are you in using the balanced food pyramid as a food guide for each meal? |
| 9 | How confident are you in consuming animal protein sources at every meal? (eggs, red meat, chicken) |
| 10 | How often do you do continuous physical activity for 30 minutes every day? |
| 11 | How confident are you in eating fruit at every meal? |
| 12 | How confident are you in washing your hands after using the bathroom? |
| 13 | How confident are you in helping clean your environment every day? |

| Name : | |
|-----------------|-------|
| School/ Class : | Age : |

| ••• | ••• | • • • • | ••• |
|-----|-----|---------|-----|

| Time<br>Eat | Dish | | | | Material name | URT | Estimate | Heavy |
|---|---|---|---|---|---|---|---|---|
| Lat | Name<br>Food | Process<br>Processing | Portion<br>(in<br>URT) | Estimate<br>(grams) | -food | | (grams) | Clean<br>(grams) |
| Morning | | | | | | | | |
| Interlude | | | | | | | | |
| Afternoon | | | | | | | | |
| nterlude | | | | | | | | |
| Evening | | | | | | | | |

| Interlude |
|-----------|

#### FOOD FREQUENCY FORM

#### SQ-FFQ (SEMI QUANTITATIVE FOOD FREQUENCY QUESTIONNARE)

| Name : |
|-----------------------|
| School/ Class : Age : |

| No | Food Names | Heavy | Portion | Freque | ency | | | Portio | on | | Flat-<br>flat<br>x/H | Heavy<br>g/H |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | rood ivallies | (g) | | х/Н | X/M | х/В | No<br>Prnh | K | S | В | | |
| Stapl | le food | | | | l | | I | 1 | I | | | |
| 1 | White rice | 200 | 1 person at the moment | | | | | | | | | |
| 2 | Yellow rice | 200 | 1 person at the moment | | | | | | | | | |
| 3 | Fried rice | 200 | 1 person at the moment | | | | | | | | | |
| 4 | Buras | 95 | 1 pc | | | | | | | | | |
| 5 | Ketupat | 110 | 1 pc | | | | | | | | | |
| 6 | White bread | 30 | 2 slices | | | | | | | | | |
| 7 | Instant noodles | 80 | 1 pack | | | | | | | | | |
| 8 | Potato | 40 | 1 pc medium | | | | | | | | | |
| Animal S | Side Dishes | L | ı | I | 1 | Г | ı | 1 | ı | 1 | | 1 |
| 9 | Beef | 35 | 1 pm today | | | | | | | | | |
| 10 | Beef liver | 50 | 1 pm today | | | | | | | | | |
| 11 | Chicken meat | 45 | 1 pm today | | | | | | | | | |

| 12 | Chicken liver | 35 | 1 pc medium | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 13 | Rabbitfish | 45 | 1/3 tail | | | | | | | | |
| 14 | Flying fish | 45 | 1/3 tail | | | | | | | | |
| 15 | Snapper | 45 | 1/3 tail | | | | | | | | |
| 16 | Skipjack tuna | 45 | 1/3 tail | | | | | | | | |
| 17 | Milkfish | 45 | 1/3 tail | | | | | | | | |
| 18 | bete-bete fish | 45 | 1 tail kcl | | | | | | | | |
| 19 | Mairo fish | 45 | 10 tail<br>kcl | | | | | | | | |
| 20 | Fish cake | 50 | 1 pm | | | | | | | | |
| 21 | Freshwater fish (tilapia fish, mas, catfish, etc.) | 45 | 1/3 tail | | | | | | | | |
| 22 | Fresh shrimp | 35 | 4 tails sdg | | | | | | | | |
| 23 | Crab | 30 | 1 tail | | | | | | | | |
| 24 | Clams/oysters | 10 | 1 pc | | | | | | | | |
| 25 | Squid | 45 | 1 tail kcl | | | | | | | | |
| 26 | Meatball | 25 | 1 seed | | | | | | | | |
| 27 | Sausage | 20 | 1 seed | | | | | | | | |
| 28 | Dried fish | 20 | 11 tails | | | | | | | | |
| 29 | Anchovy | 15 | 2 tbsp | | | | | | | | |
| 30 | Beef floss | 10 | 2 tsp | | | | | | | | |
| 31 | Egg chicken village | 40 | 1 piece | | | | | | | | |
| 32 | Chicken eggs | 55 | 1 piece | | | | | | | | |
| 33 | Duck eggs | 60 | 1 piece | | | | | | | | |
| 34 | Quail eggs | 10 | 2 pieces | | | | | | | | |
| 35 | Other | | | | | | | | | | |
| Vegetable Si | l<br>ide Dishes | <u> </u> | I | <u> </u> | <u> </u> | <u> </u> | <u> </u> | 1 | <u> </u> | <u> </u> | <u>l</u> |
| 36 | Know | 110 | 1 pm bsr | | | | | | | | |
| 37 | Tempeh | 50 | 2 pm today | | | | | | | | |
| 38 | Mung beans | 15 | 1 tbsp | | | | | | | | |
| 39 | Peanuts | 15 | 1 tbsp | | | | | | | | |
| 40 | Cashew nuts | 15 | 1 tbsp | | | | | | | | |

| 44 | Other | | |
|---------|-----------------|-----|--------------|
| 41 | | | |
| Vegetab | Vegetables | | |
| 42 | Spinach | 50 | 1 prg |
| 43 | Broccoli | 100 | 1 gls |
| 44 | Beans | 50 | 7 pcs |
| 45 | Cassava leaves | 50 | 1 prg |
| 46 | Corn | 50 | 1/3 pm |
| 47 | Mold | 15 | 1½ tbsp |
| 48 | Banana heart | 15 | 1 tbsp |
| 49 | Long beans | 50 | 3 pcs |
| 50 | Spinach | 50 | 1 prg |
| 51 | Cauliflower | 20 | 2 tbsp |
| 52 | Cabbage | 50 | 1/8 pm |
| 53 | Summer squash | 50 | 1 pm today |
| 54 | Chayote | 50 | 1 pm today |
| 55 | Cucumber | 20 | 2 slices |
| 56 | Young Jackfruit | 20 | 2 tbsp |
| 57 | Bamboo shoots | 30 | 2 tbsp |
| 58 | Mustard greens | 50 | 1 prg |
| 59 | Bean sprouts | 15 | 1 tbsp |
| 60 | Eggplant | 50 | ½ hour |
| 61 | Tomato | 25 | 1 seed |
| 62 | Carrot | 50 | ½ pcs |
| 63 | Other | | |
| Fruits | 5 | | • |
| 64 | Avocado | 50 | ½ fruit |
| 65 | Apple | 75 | ½ fruit |
| 66 | Guava | 100 | 1 pc medium |
| 67 | Orange | 150 | 1 pc medium |
| 68 | Ambarella | 100 | 1 pc medium |
| 69 | Mango | 90 | ½ pcs medium |
| 70 | Pawpaw | 110 | 1 pm today |
| 71 | Rambutan | 75 | 5 pieces |
| 72 | Watermelon | 180 | 2 pm today |

| 73 | Wine | 125 | 11 pieces | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| 74 | Pear | 85 | ½ fruit | | | | | | |
| 75 | Banana | 50 | 1 piece | | | | | | |
| 76 | Snakefruit | 80 | 1 piece | | | | | | |
| 77 | Durian | 35 | 3 seeds | | | | | | |
| 78 | Long-haired | 75 | 5 pieces | | | | | | |
| 79 | Melon | 100 | ½ pg bsr | | | | | | |
| 80 | Pineapple | 95 | ¼ pcs medium | | | | | | |
| 81 | Other | | | | | | | | |
| Drinks | & Supplements | | • | | | • | ı | | |
| 82 | Milk powder | 10 | 1 tbsp | | | | | | |
| 83 | UHT Milk | 200 | 1 gls | | | | | | |
| 84 | Soy milk | 200 | 1 gls | | | | | | |
| 85 | Milk thick sweet | 10 | 1 tbsp | | | | | | |
| 86 | Milo cans | 240 | 1 set | | | | | | |
| 87 | Milo sachet | 14 | 1 pack | | | | | | |
| 88 | Frisian flag | 190 | 1 box | | | | | | |
| 89 | Energen | 30 | 1 pack | | | | | | |
| 90 | Cheese | 10 | 1 tbsp | | | | | | |
| 91 | Ice cream | 125 | 1 cup | | | | | | |
| 92 | Ice cream stick<br>(Feast, Paddle<br>pop, etc.) | 65 | 1 pack | | | | | | |
| 93 | Signature Supplement | | 1 tablet | | | | | | |
| Snack | Food | l | <u> </u> | | l | • | I | ı | I |
| 94 | Donuts | 65 | 1 pc | | | | | | |
| 95 | Rissoles | 50 | 1 pc | | | | | | |
| 96 | Pudding | 65 | 1 pc | | | | | | |
| 97 | Brownies | 30 | 1 pc | | | | | | |
| 98 | Fried sweet potatoes | 60 | 1 pc | | | | | | |
| 98 | Fried breadfruit | 13 | 1 pc | | | | | | |
| 100 | Fried bananas | 60 | 1 pc | | | | | | |
| | | | 1 | 1 | | | | | |
| 101 | Fritters | 40 | 1 pc | | | | | | |

| 103 | Bright moon | 50 | 1 pm today |
|---|---|---|---|
| 104 | Pancakes | 40 | 1 pm today |
| 105 | Green banana | 60 | 1 pc |
| 106 | The hammer is broken | 220 | 1 mgk |
| 107 | Tella tella | 120 | 1 prg |
| 108 | The Road | 65 | 1 pc |
| 109 | Know the contents | 20 | 1 pc |
| 110 | chicken Soto | 225 | 1 mgk |
| 111 | Coto | 400 | 1 mgk |
| 112 | Meatball noodles | 370 | 1 mgk |
| 113 | Dumplings | 390 | 1 mgk |
| 114 | Mixed vegetables with the peanut sau | <sub>e</sub> 430 | 1 prg |
| 115 | Batagor | 220 | 1 prg |
| 116 | dumpling | 160 | 1 mgk |
| 117 | Titi noodles | 400 | 1 prg |
| 118 | Chicken satay | 80 | 5 tsk |
| 119 | Other | | |

## RAYMOND B. CATTELL KAREN S. CATTELL

# CFIT SKALA 3 BENTUK A

PENGGUNAAN TERBATAS HANYA OLEH PSIKOLOG



LEMBAGA PENGEMBANGAN SARANAN PENGUKURAN DAN PENDIDIKAN PSIKOLOGI FAKULTAS PSIKOLOGI - UNIVERSITAS INDONESIA 1996

#### Contoh







JANGAN MENULIS ATAU MEMBUAT CORETAN DI DALAM BUKU INI

UI - 10442 - 96

e 2 Ь d a C 3 e Ь a

(0)

Lambara Danas Banasa Carana Banaskuran dan Bandidikan Beikali

3















Contoh



1000





#### Contoh











4

#### Contoh





